CLINICAL TRIAL: NCT04902807
Title: Conception of a Diagnosis, Prognosis and Therapeutic Decision Tool for Patients With Autoimmunity and Inflammation
Acronym: ATRACTion
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-59
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Lymphoproliferative Syndrome; Autoimmune Cytopenia; Autoimmune Diseases; Autoimmune Anemia; Autoimmune Thrombocytopenia; Autoimmune Hepatitis; Autoimmune Diabetes; Autoimmune Rheumatologic Disease; Systemic Lupus Erythematosus; Juvenile Idiopathic Arthritis; Hemophagocytic Lymphohistiocytoses; EBV Lymphoproliferation; RAS-Associated Autoimmune Leucoproliferative Disease; Primary Immunodeficiency; APECED; IPEX; BENTA; Enteropathy, Autoimmune; Combined Immunodeficiency; IBD
MeSH Terms: conditions — Autoimmune Lymphoproliferative Syndrome; Autoimmune Diseases; Purpura, Thrombocytopenic, Idiopathic; Hepatitis, Autoimmune; Diabetes Mellitus, Type 1; Lupus Erythematosus, Systemic; Arthritis, Juvenile; Lymphohistiocytosis, Hemophagocytic; Primary Immunodeficiency Diseases; Polyendocrinopathies, Autoimmune; Autoimmune enteropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine and Stools
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: based on the potential for inclusion of patient's cohort followed in Necker hospital with PIDs and poly-autoimmunity related to known genetic defects. Recruitments will be made at Pediatric Rheumatology Immuno Hematology department, and paediatric Gastroenterology department (n=250).
  Collection of blood, urine and stools at inclusion and blood at 12 months consultation/ follow-up.
  Interventions: Biological: Collection of samples
- Patients' relatives (control): Brothers or sisters of the patients (n=125). Collection of blood, urine and stools at inclusion.
  Interventions: Biological: Collection of samples
- Patients with unrelated diseases (control): Recruitments will be made at the Paediatric Gastroenterology Department, in the Department of Paediatric Visceral and Urologic Surgery and the Department of Maxillofacial Surgery and Paediatric Plastic Surgery at Necker's Hospital. Participants will be included if not diagnosed PIDs and poly-autoimmunity (n=125).
  Collection of blood, urine and stools.
  Interventions: Biological: Collection of samples

INTERVENTIONS:
Biological: Collection of samples — Blood, Urine and Stool samples will be collected from the participants.

SUMMARY:
The main objective of this study is to generate diagnosis and therapeutic-decision tools through the identification of molecular causes of PIDs with autoimmunity/inflammation and the variability in disease outcome at the transcriptional level using a combination of omics signatures (transcriptomics, epigenomics, proteomics, metagenomics, metabolomics and lipidomics).

DETAILED DESCRIPTION:
Primary Immune deficiencies (PIDs) are a group of monogenic diseases related to developmental or functional dysfunction of one or several immune cell types. Individually there are rare entities, but collectively they group several thousands of patients.

Approximately 500 000 patients suffer from PIDs worldwide, making their management a true health-care concern. According to European Society for Immunodeficiencies (ESID), the age group in which PIDs is most frequently diagnosed is under 19 years of age (62%)1. PIDs are causing susceptibility to severe and life-threatening infections by common pathogens, but they also predispose to cancer and can initially manifest as autoimmune and inflammatory diseases.

Multiple mechanisms underlie the development of autoimmunity/inflammation in PIDs. Moreover, their development can be influenced by the composition of the microbiota, which shapes host metabolic and immune functions and can be modified by many environmental factors. In the last two decades a particular emphasis was given to the elucidation of the genomic mutations causing PIDs. This led to a burst of genetic diagnosis as the numbers of known monogenic causes of PIDs rose from around 200 in 2010 to more than 310 in 2017. These genomic approaches revealed that: 1) a given monogenic defect can lead to very dissimilar clinical presentations, disproving the initial concept that a monogenic defect is associated with specific clinical manifestations ; and 2) the number of cases of autosomal dominant genetic deficiencies has increased, with sometimes a partial clinical penetrance so that some relatives carrying the causal genetic variant remain asymptomatic. Hence, onset and presentation of autoimmune and inflammatory diseases in PIDs is highly unpredictable.

PIDs with autoimmunity/inflammation usually require life-long symptomatic treatments including broad immunosuppression or immunotherapies. On the long term, such treatments can have important side effects or poor efficacy and they result in high burden cost. It is therefore crucial to diagnose PIDs as early as possible in order to select the most efficient therapy based not only on clinical features as it is nowadays, but to include the underlying molecular cause of immune dysregulation.

The central goal of this project is to explain the very variable outcome of monogenic autoimmune and inflammatory diseases and to define predictive biomarkers in order to stratify patients and to optimize therapeutic choices.

ELIGIBILITY:
Inclusion Criteria for controls (patients relatives and unrelated subjects):

* Individuals aged<18 y/o.
* Individuals > 6 kg
* Individuals not affected by an immune-related disease or not affected by cancer
* Individuals whose parents have signed an enlightened consent.

Inclusion criteria for patients

* Individuals with health insurance.
* Patients treated at Necker hospital with PIDs and autoimmunity/inflammation related to known genetic defects (cytopenia, Enteropathy Inflammatory bowel disease (IBD), Systemic Lupus Erythematosus (SLE), Juvenile Idiopathic Arthritis (JIA), Familial Hemophagocytic Lymphohistiocytosis (FHL), chronic EBV infection associated (Ca-EBV) with EBV-infected T and/or Natural Killer (NK) cells and with a high risk to develop macrophage activation syndrome similar to FHL. See table below for diagnosis inclusion criteria.
* Individuals aged<18 y/o.
* Individuals > 9 kg
* Patients whose parents have signed an enlightened consent.

Exclusion Criteria:

* Intake of antibiotics within 2 weeks prior inclusion
* Absence of parent's or child consent form
* Cytotoxic cancer treatments
* antiviral treatments (HIV, hepatitis …)
* Short term life-threatening conditions
* Individuals placed under judicial protection

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with PIDs and autoimmunity/inflammation related to known and unknown genetic defects (ALPS, Cytopenia, Enteropathy-IBD, pSLE, JIA, FHL, CA-EBV, CID) and their healthy relatives (controls) will be recruited in 2 clinical services of Necker hospital: Paediatric Rhumatology Immuno Hematology department Department, and paediatric Paediatric Gastroenterology department Department.
  Unrelated controls will be recruited in the Paediatric Rhumatology Immuno Hematology Department, the Paediatric Gastroenterology Department,also be recruited in the Department of Paediatric Visceral and Urologic Surgery and the Department of Maxillofacial Surgery and Paediatric Plastic Surgery within patients hospitalised for a surgery and not affected by an immune-related disease or a cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Generate a diagnosis and therapeutic-decision tools | 5 years
  Identification of molecular causes of PIDs with autoimmunity/inflammation and the variability in disease outcome at the transcriptional level using a combination of omics signatures (transcriptomic, epigenomics, proteomic, metagenomic, metabolomics and lipidomics).

SECONDARY OUTCOMES:
1- Development of an atlas of molecular interactions leading to autoimmunity and inflammation | 5 years
  Research tool integrating transcriptomic, proteomic, epigenetic, metabolomic and lipidomics data of pediatric affected patients as well as healthy pediatric individuals This atlas will be available widely to the public and private research community.
2 - To develop an artificial intelligent online application | 5 years
  The decision support tool will be interoperable with any clinical information system and will be clinically validated.
3- Ancillary study (pilot study) | 5 years
  i. Validation of candidate biomarkers associated to diagnosis and prognosis of Juvenile Idiopathic Arthritis patients ; ii. Definition of a specific clinical outcome and early quantification of the performance of a diagnostic decision tool based on omics signatures (proof of concept)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Rieux-Laucat, Principal Investigator — Institut Imagine
Locations (1):
- hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of the research study — https://atraction.institutimagine.org/en